CLINICAL TRIAL: NCT02726204
Title: Evaluation of a Wearable Exoskeleton for Functional Arm Training (CAREX)
Brief Title: Evaluation of a Wearable Exoskeleton for Functional Arm Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 15-00402
Record Dates: First submitted 2016-03-17; First posted 2016-04-01 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Stroke; Post-Stroke Hemiparesis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Subjects (Active Comparator): Seven healthy patients will serve as controls based on preliminary data in healthy volunteers using CAREX with gravity elimination alone versus gravity elimination plus path assistance.
  Interventions: Other: Gravity Elimination Alone; Other: Path Assistance Alone; Other: Path Assistance and Gravity Elimination
- Chronic Post Stroke Right Side Hemiparesis (Active Comparator): Radiologically verified unilateral stroke patients with at least 4 months previously.
  Interventions: Other: Gravity Elimination Alone; Other: Path Assistance Alone; Other: Path Assistance and Gravity Elimination

INTERVENTIONS:
Other: Gravity Elimination Alone — CAREX will compensate for the gravity of the subject's arm, i.e. subject can move their arm to a specific position and relax all the arm muscles, CAREX will hold the arm in that configuration
Other: Path Assistance Alone — CAREX will push subject's arm to a pre-specified path. If the arm is not in the path, CAREX will generate some force that is proportional to the distance between the hand and the path. The subject will feel like having a spring connected between his hand and the path
Other: Path Assistance and Gravity Elimination

SUMMARY:
The purpose of this study is to investigate how the cable-driven arm exoskeleton (CAREX) can assist task performance during 3D arm movement tasks under various experimental conditions in healthy individuals and patients with stroke. This study is designed to test motor learning with the robotic rehabilitative device CAREX under three conditions in healthy subjects and subjects with post-stroke hemiparesis.

ELIGIBILITY:
Inclusion Criteria for stroke population:

* Radiologically verified unilateral stroke at least 4 months previously.
* Right-handed subjects with or without right hemiparesis (as robot is built for right arm alone).
* Preserved passive range of motion at all upper limb joints.
* Spasticity <3 on the modified Ashworth Scale (MAS).
* Ability to follow study instructions and likely to complete the protocol; ability to comply with the protocol as assessed by the investigator; must be English speaking since the assessments are in English.

Exclusion Criteria for stroke population.

* History of surgery or other significant injury to either upper extremity causing mechanical limitations that preclude task performance.
* Previous neurological illness such as head trauma, prior stroke ( as we are recruiting subjects with first unilateral stroke), epilepsy, or demyelinating disease.
* Complicating medical problems such as uncontrolled hypertension, diabetes with signs of polyneuropathy, severe renal, cardiac or pulmonary disease, or evidence of other concurrent neurologic or orthopedic conditions precluding the subject from complying with the study protocol.
* Severe upper extremity spasticity suggested by an Ashworth score of >3 at any joint, or restriction of full passive range of motion.
* Evidence of alcohol, drug abuse or other relevant neuropsychiatric condition such as psychotic illness or severe depression.

Inclusion Criteria for control population.

* No previous stroke or any other previous neurological injury.
* Right-handed subjects without any weakness or hemiparesis (as robot is built for right arm alone).
* Preserved passive and active range of motion at all upper limb joints.
* No increase in muscle tone in response to passive range of motion. A score of zero on Ashworth Scale (MAS).
* Able to achieve full score on upper extremity Fugl-Meyer Scale (66/66)
* Ability to follow study instructions and likely to complete the protocol; ability to comply with the protocol as assessed by the investigator; must be English speaking since the assessments are in English.

Exclusion Criteria for control population.

* History of surgery or other significant injury to either upper extremity causing mechanical limitations that preclude task performance.
* Previous neurological illness such as head trauma, prior stroke, epilepsy, or demyelinating disease.
* Complicating medical problems such as uncontrolled hypertension, diabetes with signs of polyneuropathy, severe renal, cardiac or pulmonary disease, or evidence of other concurrent neurologic or orthopedic conditions precluding the subject from complying with the study protocol.
* Any condition or situation that, in the investigator's opinion, may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
* Severe upper extremity spasticity suggested by an Ashworth score of >3 at any joint, or restriction of full passive range of motion.
* Evidence of alcohol, drug abuse or other relevant neuropsychiatric condition such as psychotic illness or severe depression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Passive range of motion measured by goniometry | 1 Day
Active range of motion measured by goniometry | 1 Day
Upper extremity motor impairment measured by performance on the 33 tasks of the Fugl-Meyer Scale (FMS) | 1 Day
Spasticity measured by the Modified Ashworth Scale (MAS) | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Raghavan, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States